CLINICAL TRIAL: NCT02565680
Title: Glucocorticoids Associated With Antihistamines Versus Antihistamines Randomized Double Blinded for the Management of Acute Urticaria in Emergency
Brief Title: Glucocorticoids With Antihistamines Versus Antihistamines in Acute Urticaria in Emergency
Acronym: CAHISU
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11 221 02
Record Dates: First submitted 2014-07-22; First posted 2015-10-01 (Estimated); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Acute Urticaria
Keywords: acute urticaria; glucocorticoids; antihistamines; prurit; itch score; rash
MeSH Terms: conditions — Exanthema | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): tablets of Xyzall 5mg/ day during 5 days + placebo 40mg/ day during 4 days
  Interventions: Drug: placebo
- prednisone (Experimental): tablets of Xyzall 5 mg/j during 5 days + prednisone 40 mg/ day during 4 days
  Interventions: Drug: prednisone

INTERVENTIONS:
Drug: placebo — Xyzall 5mg during 5 days + placebo 40mg during 4 days
  Arms: placebo
Drug: prednisone — Xyzall 5mg during 5 days + prednisone 40mg during 4 days
  Arms: prednisone

SUMMARY:
Acute urticaria is common and affected 12% of population. 400 patients come in department emergency of Toulouse each year and there aren't many studies in literature which evaluate the glucocorticoids treatment. The standard treatment of urticaria is antihistamines H1, but glucocorticoids treatment administered orally for short course would permit to increase quickly acute urticaria uncomplicated. Clinical trial, prospective randomized double blinded of adults with acute urticaria less 24 hours duration and no take treatment urticaria before.

DETAILED DESCRIPTION:
Acute urticaria is common and affected 12% of population. 400 patients come in department emergency of Toulouse each year and there aren't many studies in literature which evaluate the glucocorticoids treatment. Acute urticaria is pruritic and incapacitating for daily life. The standard treatment of urticaria is antihistamines H1, but glucocorticoids treatment administered orally for short course would permit to increase quickly acute urticaria uncomplicated. Clinical trial, prospective randomized double blinded of adults with acute urticaria less 24 hours duration and no take treatment urticaria before. One group randomized received 40mg of cortancyl and 1 pill of citerizine and another group randomized received 1 pill citerizine and placebo like cortancyl. Pharmacy hospital takes care of randomization. Pruritus evaluated with icth score and rash evaluated with nine rule of Wallace, the patient is evaluated in T0, one hour after and contacted by telephone at J2, J5, J15, J 21 itch score, Wallace extension, observance, side effects are asked him.

ELIGIBILITY:
Inclusion Criteria:

* adults
* urticaria rash no more 24 h duration and no take treatment for urticaria

Exclusion Criteria:

* patients were presented severe anaphylaxis or taken antihistamines or glucocorticoids within 5 days of arrival at ED,
* severe infection
* pregnancy
* patients BPCO
* diabetics
* allergy corticosteroids
* refusal to comply
* participate an other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To compare treatment with prednisone and antihistamines versus antihistamines placebo to out acute urticaria in 48 hours | 48 hours
  To compare treatment with prednisone and antihistamines versus antihistamines placebo to out acute urticaria in 48 hours using the itch score

SECONDARY OUTCOMES:
Evolution of intensity pruritus, angioedema and rash with nine rule of Wallace | 21 days
  Evolution of intensity pruritus at T0 and T1, J2, J5, J15, J21 and angioedema and rash at T1, J2, J5, J15 and J21 comparing at T0 with nine rule of Wallace
The necessary time to decrease pruritus and rash | 21 days
  The necessary time to decrease pruritus and rash
The frequency of side-effects in either treatment group in 21 days | 21 days
  The frequency of side-effects in either treatment group in 21 days
Recidive of urticaria | 21 days
  The recidive of urticaria
The observance treatment | 21 days
  Observance treatment

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Barniol, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

REFERENCES:
- [Result] Barniol C, Dehours E, Mallet J, Houze-Cerfon CH, Lauque D, Charpentier S. Levocetirizine and Prednisone Are Not Superior to Levocetirizine Alone for the Treatment of Acute Urticaria: A Randomized Double-Blind Clinical Trial. Ann Emerg Med. 2018 Jan;71(1):125-131.e1. doi: 10.1016/j.annemergmed.2017.03.006. Epub 2017 May 3. PMID 28476259